CLINICAL TRIAL: NCT06247709
Title: Evaluation of KLHL14 Expression as a Prognostic Factor of PitNET Invasiveness
Brief Title: KLHL14 Expression as Predicting Factor of Invasiveness in pitNET
Status: Completed | Type: Observational
Sponsor: Federico II University (Other)
Collaborators: University of Teramo (Other)
Responsible Party: Principal Investigator, Domenico Solari, Associate Professor of Neurosurgery, Federico II University
Other Study IDs: 17-1-j
Record Dates: First submitted 2024-01-12; First posted 2024-02-08 (Actual); Last update posted 2024-02-08 (Actual); Status verified 2024-02

CONDITIONS: Invasiveness, Neoplasm
MeSH Terms: conditions — Neoplasm Invasiveness

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — Tissue samples of pituitary adenoma cell, taken off during surgery
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Cases: All patients undergone surgery for the removal of a pituitary adenoma. Tissue samples of these cases were sent to biochemical essay to measure the expression and localisation of KLHL14.
  Interventions: Other: Immunohistochemical expression in pitNET cells of KLHL14

INTERVENTIONS:
Other: Immunohistochemical expression in pitNET cells of KLHL14 — Lab essay evaluating the expression of KLHL 14

SUMMARY:
OBJECTIVE: The objective of this study is to evaluate the correlation between KLHL14 expression and its cytoplasm-nuclear localisation and pituitary adenomas biological behaviour with particular focus on its role in epithelial mesenchymal transition and invasion of para and suprasellar regions.

This is a multicenter and multidisciplinary study, with the involvement of the Departments of Neurosurgery of the University of Naples Federico II and the Department of Biosciences of the University of Teramo.

DETAILED DESCRIPTION:
The investigators would like to analyse the possible correlations between the expression, the cytoplasm-nuclear localisation and the activity of the protein KLHL14 and pituitary adenomas biological behaviour with particular focus on its role in epithelial mesenchymal transition and invasion of para and suprasellar regions. This study will be conducted on biological sample collected during surgery and primary cellular line derived from those samples.

Patients refer to neurosurgery for the detection of pituitary adenomas with various presenting symptoms that can be correlated to hormone production or to mass effect produced by the lesion on the optic apparatus or on the oculomotor nerves after invasion of the cavernous sinus. All patients undergo an ophthalmological clinical examination to define the presence of visual alteration and endocrinological assessment to determine eventual hormone hypersecretion. Finally, radiological exams, as magnetic resonance of the sellar region, are performed on patients to evaluate the extension of the pathology, its relationship to the surrounding neurovascular structures and therefore guide neurosurgical resection which is typically performed via an endoscopic endonasal transsphenoidal approach. Except for prolactin secreting pituitary adenomas, for which medical therapy with dopaminergic agonists is a viable approach, surgery with adenoma resection represent the gold standard for treatment.

ELIGIBILITY:
INCLUSION CRITERIA:

* Adult men or women (age 18-70)
* Patients affected by nonfunctioning pituitary adenomas.

EXCLUSION CRITERIA:

* Prisoners
* Pregnant women
* Patient under 18 years
* Patients without capacity of discernment.

Ages: 18 Years to 70 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: All consecutive cases of radiologically invasive pitNET undergoing tumor removal
Sampling Method: Non-Probability Sample
Enrollment: 12 (Actual)
Dates: Start 2023-03-12 (Actual); Primary Completion 2023-10-31 (Actual); Study Completion 2023-12-17 (Actual)

PRIMARY OUTCOMES:
Invasiveness degree | Invasiveness degree will be determined at the time of surgery
  The expression of KLHL14 in invasive pituitary adenomas

CONTACTS AND LOCATIONS:
Overall Officials: Barbara Barboni, PhD, Principal Investigator — University of Teramo
Locations (1):
- Federico II university, Napoli, Italy

IPD SHARING:
Plan to Share IPD: No